CLINICAL TRIAL: NCT06299332
Title: Safety and Efficacy of Bi-Polar Radiofrequency for the Treatment of Erectile Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: InMode MD Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DO611503A
Record Dates: First submitted 2023-11-27; First posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2023-11

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Intervention Model Description: Prospective, open-label clinical study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Device Treatment (Experimental): Eligible subjects will receive 6 weekly treatments with the Forma Applicator according to the study protocol and will return for two follow up visits 1- and 3-months post treatment. Two further telephone feedback checks will be carried out 6 months and 12 months following the last treatment visit.
  Interventions: Device: Device treatment

INTERVENTIONS:
Device: Device treatment — 20 heterosexual males clinically diagnosed with Erectile Dysfunction will receive 6 weekly treatments with the Forma Applicator according to the study protocol and will return for two follow up visits 1- and 3-months post treatment. Two further telephone feedback checks will be carried out 6 months and 12 months following the last treatment visit

SUMMARY:
The goal of this prospective pilot study is to learn about the Safety and Efficacy of Radiofrequency (RF) for the Treatment of Erectile Dysfunction. This research study is trying to determine if RF therapy is safe and effective in patients with symptoms of erectile dysfunction (ED).

ELIGIBILITY:
Inclusion Criteria:

1. Adult male between ≥40 and ≤80 years of age
2. Subjects with a history of self-reported erectile dysfunction lasting for over 6 months and not more than 5 years.
3. The subject is PDE5i responsive, meaning he is able to achieve and maintain an erection under the effect of the maximal dosage of PDE5i
4. The subject has been in a stable heterosexual relationship for over 3 months prior to enrollment.
5. A minimum of 4 sexual attempts during the last two weeks prior to enrollment.
6. Abstinence from taking PDE5 for two weeks (washout) after enrolment and 2 weeks before each follow up visit/call.
7. IIEF-EF score between 11 and 25.
8. Testosterone level 300-1000 mg/dL within 1 month prior to the enrollment/baseline.
9. A1C level ≤ 8.5% within 1 month prior to enrollemnt/baseline.
10. Subject has at EHS score ≥ 1 (natural tumescence during sexual stimulation).
11. The subjects should understand the information provided about the investigative nature of the treatment, possible benefits and side effects, and are willing to sign the Informed Consent Form
12. If the FirmTech Ring is provided, the participants must be willing to use the ring according to the instructions.
13. The subjects should be willing to comply with the study procedure and schedule, including follow up visits.
14. Agreement/ability to abstain from erectile dysfunction medications or any device treatments for the duration of the study, i.e., the time between the treatment visit and the final study visit.

Exclusion Criteria:

1. Evidence of co-existing Neurological disease or other systemic disease conditions such as Alzheimer or Parkinson disease which affects erectile function (at the discretion of the investigator)
2. History of radical prostatectomy or extensive pelvic surgery ever
3. Psychiatric diagnosis or medications such as antidepressants which affects erectile function or any other medications at the discretion of the investigator.
4. Anatomical malformation of the penis, including Peyronie's disease.
5. Testosterone level <300 or >1000 ng/dL within 1 month prior to enrollment.
6. Diabetes type I
7. Diabetes Type II with A1C level > 8.5% within 1 month prior to enrollment.
8. Unwillingness to abstain from systemic medications known to cause ED for the study duration.
9. Internal defibrillator, pacemaker or any other implanted electrical device anywhere in the body
10. Permanent metal implant in the treatment area
11. Any surgery in the treatment area in the last 3 months
12. Current or history of skin cancer, or current condition of any other type of cancer, or pre-malignant moles in the facial area
13. Impaired immune system due to immunosuppressive diseases such as AIDS and HIV, or use of immunosuppressive medications
14. Patients with history of diseases stimulated by heat, such as recurrent Herpes Simplex in the treatment area, may be treated only following a prophylactic regimen.
15. Poorly controlled endocrine disorders, such as diabetes, thyroid dysfunction
16. Any active condition in the treatment area, such as but not limited to open sores, psoriasis, eczema, vitiligo, herpes and rash.
17. History of skin disorders, keloids, abnormal wound healing, as well as very dry and fragile skin
18. Severe concurrent conditions, such as cardiac disorders, sensory disturbances.
19. Use of Isotretinoin (Accutane®) within 30 days prior to treatment.
20. Participation in another study within 30 days prior to screening.

    -

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 20 heterosexual males clinically diagnosed with Erectile Dysfunction
Enrollment: 20 (Estimated)
Dates: Start 2023-06-23 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Change in ED symptoms, following the RF treatment | 3 months
  Change in ED symptoms, following the RF treatment measured by THE INTERNATIONAL INDEX OF ERECTILE FUNCTION - ERECTILE FUNCTION (IIEF-EF) questionnaire score.
  The IIEF-5 score is the sum of the ordinal responses to the 5 items.(1 to 5 ) 22-25: No erectile dysfunction 17-21: Mild erectile dysfunction 12-16: Mild to moderate erectile dysfunction 8-11: Moderate erectile dysfunction 5-7: Severe erectile dysfunction

SECONDARY OUTCOMES:
Change in sexual activity leading to optimal penetration | 3 months
  Change in sexual activity leading to optimal penetration measured by SEP- Sexual Encounter Profile questionnaire. The SEP questionnaire consists of 5 items addressing the sexual events and subject experiences when attempting intercourse. Efficacy of RF treatment evaluated using the change in percentage of "yes" responses to Sexual Encounter Profile (SEP) Questions 2 and 3
Evaluate efficacy of the RF treatment for erectile function | 3 months
  Proportion of subject responses to Global Assessment Questionnaire (GAQ) consisting of 2 questions (Yes or No): Question 1 'Has the treatment you have been taking improved your erectile function?' and if necessary, Question 2 'If yes, has the treatment improved your ability to engage in sexual activity?'.
Evaluate efficacy of the RF treatment for erectile function | 6 months
  Proportion of subject responses to Global Assessment Questionnaire (GAQ) consisting of 2 questions (Yes or No): Question 1 'Has the treatment you have been taking improved your erectile function?' and if necessary, Question 2 'If yes, has the treatment improved your ability to engage in sexual activity?'.
Evaluate efficacy of the RF treatment for erectile function | 12 months
  Proportion of subject responses to Global Assessment Questionnaire (GAQ) consisting of 2 questions (Yes or No): Question 1 'Has the treatment you have been taking improved your erectile function?' and if necessary, Question 2 'If yes, has the treatment improved your ability to engage in sexual activity?'.
Evaluate efficacy of the RF treatment for hardness of erection | 3 months
  To assess the effectiveness of RF treatment for erectile dysfunction with the Erectile Hardness Score (EHS) questionnaire The Erection Hardness Score is a self-reported tool that measures the hardness of an erection.
  It involves a scale report from 0 to 4, 4 being the best quality of erection.

OTHER OUTCOMES:
Measuring pain level during the procedure | During the procedure
  NPRS is a unidimensional measure of pain intensity in adults. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").

CONTACTS AND LOCATIONS:
Overall Officials: Robert Valenzuela, MD, Principal Investigator; Lanna Cheuck, MD, Principal Investigator
Locations (2):
- United States (2):
  - LC Medical 140 W 58th St, Suite A New York, NY 10019, New York, New York
  - Washington Heights Urology, New York, New York

IPD SHARING:
Plan to Share IPD: No